CLINICAL TRIAL: NCT00136474
Title: A Randomized Phase II Trial of Amifostine for Head and Neck Irradiation in Lymphoma
Brief Title: Amifostine for Head and Neck Irradiation in Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); MedImmune LLC (Industry)
Responsible Party: Andrea K. Ng, MD, Dana-Farber Cancer Institute/Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-292
Record Dates: First submitted 2005-08-25; First posted 2005-08-29 (Estimated); Last update posted 2009-11-02 (Estimated); Status verified 2009-10

CONDITIONS: Lymphoma; Hodgkin's Disease; Non-Hodgkin's Lymphoma
Keywords: Lymphoma; Radiation therapy; Amifostine
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin | interventions — Amifostine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Amifostine plus radiation therapy
  Interventions: Drug: Amifostine; Radiation: Radiation Therapy
- Group 2 (Active Comparator): Radiation therapy alone
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Amifostine — Given 30-60 minutes prior to daily radiation therapy
  Arms: Group 1
Radiation: Radiation Therapy — Daily radiation therapy

SUMMARY:
The purpose of this study is determine the effects (good and bad) amifostine has on radiation-induced side effects of lymphoma treatment.

DETAILED DESCRIPTION:
Patients will be randomized into one of two study groups. One study group will receive amifostine prior to daily radiation therapy and the other group will receive radiation therapy alone.

Amifostine will be administered 30-60 minutes prior to radiation treatment. Vital signs will be monitored 5 minutes and 15 minutes after amifostine injection as well as immediately following radiation treatment.

Patients will also complete a quality-of-life questionnaire on the first and last day of radiation treatment. Follow-up questionnaires will be done at follow-up visits 1 month, 3 months, 6 months, 12 months, 18 months and 24 months after completion of radiation therapy.

Patients will be removed from the study if they develop an allergic reaction to amifostine.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 35 years or older
* Histologically confirmed Hodgkin's disease or non-Hodgkin's lymphoma receiving radiation therapy to the head and neck area.
* Involvement of one or more of the following sites: cervical node, supraclavicular node, pre-auricular node, submental node, any salivary glands, any parts of the oral cavity, or any parts of the oropharynx.

Exclusion Criteria:

* Prior history of head and neck malignancies
* Prior radiation therapy to the head and neck region
* Patients with stage I Hodgkin's disease receiving radiation therapy alone
* Pregnant or lactating women
* Myocardial infarction within the 6 months of enrollment
* Clinically evident pulmonary insufficiency, except for patients with exertional dyspnea related to chest tumor itself.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2003-05; Primary Completion 2005-05 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the effectiveness of amifostine in reducing acute and chronic radiation-induced side effects | 2 years

SECONDARY OUTCOMES:
To determine the quality-of-life of patients receiving radiation therapy and amifostine
to determine the safety of amifostine | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Andrea K. Ng, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts